CLINICAL TRIAL: NCT00004258
Title: A Phase I Trial of EMD 121974 in Patients With Advanced or Metastatic Cancer
Brief Title: EMD 121974 in Treating Patients With Locally Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: George Sledge, MD/ Principal Investigator, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9909-40; T99-0076; IUMC-9909-40; NCI-T99-0076
Record Dates: First submitted 2000-01-28; First posted 2004-07-26 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous/Nonmalignant Condition; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; monoclonal gammopathy of undetermined significance; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage III multiple myeloma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; small intestine lymphoma; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; polycythemia vera; essential thrombocythemia; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; prolymphocytic leukemia; primary systemic amyloidosis; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; chronic idiopathic myelofibrosis; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Hodgkin Disease; Monoclonal Gammopathy of Undetermined Significance; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Blast Crisis; Polycythemia Vera; Thrombocythemia, Essential; Leukemia, Hairy Cell; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Primary Myelofibrosis; Lymphoma, B-Cell, Marginal Zone | interventions — Cilengitide

INTERVENTIONS:
Drug: cilengitide — dose escalation of cilengitide

SUMMARY:
RATIONALE: EMD 121974 may stop the growth of cancer by stopping blood flow to the tumor.

PURPOSE: Phase I trial to study the effectiveness of EMD 121974 in treating patients who have locally advanced or metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and tolerability of EMD 121974 in patients with advanced or metastatic cancer. II. Correlate various surrogate markers of antiangiogenic activity with EMD 121974 therapy including magnetic resonance imaging and PET scans, serum assays for various angiogenic and antiangiogenic factors, serum and urine markers of calcium metabolism, and tumor biopsies.

OUTLINE: This is a dose-escalation study. Patients receive EMD 121974 IV over 1 hour twice weekly for 4 weeks. Treatment continues for an additional course in the absence of unacceptable toxicity. Patients with stable or responding disease may continue therapy indefinitely past the 2 courses until disease progression. Cohorts of 3-6 patients receive escalating doses of EMD 121974 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicities. Patients are followed every 3 months for the first year, and then every 4 months thereafter until disease progression.

PROJECTED ACCRUAL: A total of 31-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed locally advanced or metastatic cancer that is considered incurable and for which no standard curative therapy exists No primary CNS malignancies Measurable evidence of residual, recurrent, or metastatic disease No prior CNS metastases with residual abnormal findings on neuroradiologic studies Prior CNS metastases allowed provided at least 6 months from definitive therapy and a normal CT or MRI of the brain

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Hemoglobin at least 9 mg/dL (may be post transfusion) Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal SGOT/SGPT no greater than 2.5 times upper limit of normal PT/PTT normal Renal: Creatinine no greater than 1.5 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active infection requiring parenteral antibiotics No documented abnormal CNS exam with seizure disorder or major neuropsychiatric problems

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 2 weeks since prior hematopoietic growth factor or cytokine therapy and recovered No concurrent immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy (at least 6 weeks since prior nitrosoureas or mitomycin) and recovered No concurrent chemotherapy Endocrine therapy: No concurrent corticosteroids except for steroid replacement therapy or chronic low dose (no greater than 10 mg/day oral prednisone) therapy for nonmalignant conditions No concurrent hormonal therapy except oral contraceptives or hormonal replacement therapy Radiotherapy: At least 2 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: At least 2 weeks since prior surgery and recovered Other: At least 4 weeks since other prior investigational drugs No concurrent oral or parenteral anticoagulants except anticoagulants for central venous catheters including low dose warfarin (1-2 mg/day) and/or heparin No concurrent oral COX-2 specific inhibitors (e.g., celecoxib or rofecoxib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1999-12; Primary Completion 2001-08 (Actual); Study Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of escalating doses of twice weekly EMD 121974 in patients with cancer. | enrollement through termination

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Gordon, MD, Study Chair — Virginia G. Piper Cancer Center at Scottsdale Healthcare - Shea
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States